CLINICAL TRIAL: NCT02866253
Title: Dehydroepiandrosterone (DHEA)Supplementations Pre-IVF Cycles Improve the Outcome of Diminished Ovarian Reserve（DOR）Patients by the Increased Level of BMP-15(Bone Morphogenetic Protein 15) in Follicular Micro-environment
Brief Title: Dehydroepiandrosterone (DHEA)Supplementation Pre-IVF(In Vitro Fertilization) Cycles
Acronym: IVF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShangHaiJiAi-05
Record Dates: First submitted 2016-08-10; First posted 2016-08-15 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2016-08

CONDITIONS: Infertility
Keywords: Dehydroepiandrosterone（DHEA）; DOR（Diminished Ovarian Reserve); IVF(In vitro fertilization); BMP-15(Bone Morphogenetic Protein 15)
MeSH Terms: conditions — Infertility | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHEA Group (Experimental): DHEA 25mg t.i.d. for more than 12weeks
  Interventions: Drug: DHEA
- Control Group (No Intervention): patients without any DHEA

INTERVENTIONS:
Drug: DHEA — Interventional patients should take DHEA 25mg tid 12weeks before enter the IVF cycle.
  Other Names: Dehydroepiandrosterone
  Arms: DHEA Group

SUMMARY:
The purpose of this study is to compare the effect of pre-IVF cycles treatment with and without DHEA(Dehydroepiandrosterone) on the ovarian reserve markers, the number of oocytes obtained and IVF(in vitro fertilization) outcomes of DOR(diminished ovarian reserve) patients and the expression of BMP-15(bone morphogenetic protein 15),GDF-9（growth differentiation factor 9) and IGF-I(insulin-like growth factors-1) in follicular fluid.

DETAILED DESCRIPTION:
78 patients were enrolled according to the inclusion criterion. They were randomized into two groups, 40 were in DHEA group and 38 were in control group. The DHEA group received DHEA (Lab Hercules™) 25mg three times a day continuing more than 12 weeks prior to the start of IVF treatment till the day of egg collection and the control group got without any DHEA treatment. All of the IVF women patients were given CC(clomifene citrate)+HMG(human menopausal gonadotropin) protocol for controlled ovarian hyperstimulation. Hormonal profile including E2(estradiol),FSH(follicle-stimulating hormone) ,P(progesterone) ,LH (luteinizing hormone),T(testosterone),AFC(antral follicle account),serum and follicle AMH(anti-Mullerian hormone)levels will be repeated in follicular phase (D2 or 3) of cycle followed by an IVF treatment using CC+HMG protocol based on our standard departmental regimen. Improvement of ovarian reserve markers would be assessed by the change in serum and follicle AMH levels. Cycle characteristics including the dose of gonadotrophins use, duration of stimulation, number of oocytes obtained, number of fertilized embryos and good quality embryos will be recorded and follicular fluid will be saved for the test of DHEA-S(Dehydroepiandrosterone sulfate) and IGF-I. BMP-15 and GDF-9 expression in the follicular fluid were detected with western blot.

ELIGIBILITY:
Inclusion Criteria:

* Patients with antral follicle count <5 or AMH<1.1ng/ml and a previous poor ovarian reserve (POR)(</= 3 oocytes with a conventional stimulation protocol using at least 150 IU FSH per day,at least two episodes)

Exclusion Criteria:

* Patients with polycystic ovary or polycystic ovary syndrome, patients who had previous chemotherapy, pelvic irradiation or ovarian surgery and patients on hormonal supplementation for any indication at the time of recruitment (e.g. estrogen, testosterone or DHEA).

Ages: 25 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Implantation rate | 6 months
  Implantation status was identified by the presence of a fetal heart beat detected with an ultrasound scan at 5 weeks after embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Xi Sun, PHD, Study Chair — ShangHai Ji Ai Genetics & IVF Institute

IPD SHARING:
Plan to Share IPD: No